CLINICAL TRIAL: NCT07060144
Title: Cognitive Processing Therapy (CPT) for Perinatal Posttraumatic Stress Disorder (PTSD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Erin Richardson, Advanced Practice Nurse, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00006641
Record Dates: First submitted 2025-06-24; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Pregnancy
Keywords: PTSD; pregnancy; cognitive processing therapy; psychotherapy; trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular CPT (Experimental): Standard-model Cognitive Processing Therapy (CPT) - one 60-min session per week for 12 weeks total
  Interventions: Behavioral: Regular CPT
- mCPT (Experimental): Massed CPT - two 60-min sessions each day for 5 consecutive days (10 sessions total)
  Interventions: Behavioral: Massed CPT

INTERVENTIONS:
Behavioral: Regular CPT — Standard-model Cognitive Processing Therapy (CPT) - one 60-min session per week for 12 weeks total
  Arms: Regular CPT
Behavioral: Massed CPT — Massed CPT - two 60-min sessions each day for 5 consecutive days (10 sessions total)
  Arms: mCPT

SUMMARY:
Pregnant women with a primary diagnosis of posttraumatic stress disorder (PTSD) (PTSD Checklist for DSM-5 (PCL-5) score > 33) will be randomized to receive conventional cognitive processing therapy (CPT) (60-min session once/week for 12 weeks) or massed CPT (mCPT) (an intensive schedule of 12 60-min sessions over 5 days, approximately 2-3 sessions per day) via telemedicine, for treatment of PTSD. The research aims will be three-fold: (1) Evaluate the relative efficacy and tolerability of CPT vs. mCPT for treatment of perinatal PTSD and depression; (2) Determine the effect of CPT upon maternal-infant attachment and interaction; (3) Collect pilot data of obstetric and neonatal outcomes among those receiving the two CPT delivery schedules.

ELIGIBILITY:
Inclusion Criteria:

* Female, ages 18-46, Pregnant (< 25 weeks), able to read and write in English, History of at least 1 criterion A trauma, Primary diagnosis of PTSD (confirmed by SCID), Psychotropic medications must be stable with no changes ≥ 2 weeks (≥ 6 weeks for fluoxetine), and no medication changes can be made during the course of therapy

Exclusion Criteria:

* Not currently pregnant, Diagnosis of bipolar disorder, psychotic disorders, Suicidal ideation with plan or intent, Substance use disorder, Regular benzodiazepine use (> 4x weekly)

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Baseline, then at 1 week, 4 weeks, 8 weeks, 12 weeks, and 16 weeks following initiation of treatment in both the mCPT and traditional CPT groups
  PTSD Checklist for DSM-5 (PCL-5) will be used to collect information on PTSD symptoms. The PCL-5 for DSM-5 is a 20-item self-report measure. Higher scores reflect greater PTSD severity. Scoring is based on how much the patient has been bothered by the symptoms on a scale from "0 = not at all" to "4 = extremely." PCL-5 total symptom severity scores range from 0 to 80 with higher scores indicating greater PTSD severity. PCL-5 Monthly will be collected at Visit 1, and the PCL-5 weekly will be collected at 1 week, 4 weeks, 8 weeks, 12 weeks, and 16 weeks following initiation of treatment in both groups.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline, then at 1 week, 4 weeks, 8 weeks, 12 weeks, and 16 weeks following initiation of treatment in both the mCPT and traditional CPT groups
  The Patient Health Questionnaire-9 (PHQ-9) is used for screening, diagnosing, monitoring, and measuring the severity of depression. Nine questions each scored from 0 (Not at all) to 3 (Nearly every day). Total score ranging from 0 to 27, with higher scores indicating more severe depression: 1 - 4: Minimal or no depression, 5 - 9: Mild depression, 10 - 14: Moderate depression, 15 - 19: Moderately severe depression, and 20 - 27: Severe depression
Prenatal Attachment Inventory (PAI) | Baseline
  The Prenatal Attachment Inventory (PAI) is a 21-item questionnaire designed to assess a pregnant woman's thoughts, feelings, and experiences related to her unborn child and her level of attachment to the fetus. It uses a 4-point Likert scale for each item (4 = almost always; 3 = often; 2 = sometimes, 1 = almost never), with scores ranging from 21 to 84, where higher scores indicate a stronger prenatal attachment.
Maternal Attachment Inventory (MAI) | Once within 1-90 days following participant's delivery (i.e once within 3 months postpartum)
  The Maternal Attachment Inventory (MAI) is a 26-item, self-report questionnaire used to assess the emotional bond between a mother and her infant. It measures maternal feelings and behaviors that reflect affection and love for the baby. Higher scores on the MAI indicate a stronger maternal attachment. The scale utilizes a four-point Likert scale for responses (4 = almost always; 3 = often; 2 = sometimes, 1 = almost never), and the total score ranges from 26 to 104.
Infant CARE-Index (CARE-Index) | Once within 1-90 days following participant's delivery (i.e once within 3 months postpartum)
  The Infant CARE-Index assesses parent-infant interaction. It is a videotaped 3-5 minute free-play observation in which the adult is asked 'to play with your child as you usually would'. Gives an assessment of the best of their potential interaction at times of low stress, i.e ideal functioning, but the scores are highly correlated with attachment. The Infant CARE-Index (ICI) is unique because it can be used from birth to 15 months and in multiple locations. The videotapes are coded by reliable coders who are blind to all information about the dyad. Based on directions in the manual, the ICI yields: Adult scores on sensitivity, control, and unresponsiveness; Infant scores on cooperation, compulsivity, difficultness, and passivity. A dyadic synchrony indicative of the degree of risk to the child's future development.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Richardson, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Dell Medical School, Department of Psychiatry, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No